CLINICAL TRIAL: NCT06545864
Title: In Hospital Clinical Outcomes and Short Term Follow up of Systemic Thrombolysis Versus Catheter Directed Management for the Treatment of Acute Intermediate-high Pulmonary Embolism
Brief Title: Systemic Thrombolysis Versus Catheter Directed Management for Acute Intermediate-high Pulmonary Embolism
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam J William, Principal Investigator, Assiut University
Other Study IDs: 123456@qerty
Record Dates: First submitted 2024-07-29; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Acute Pulmonary Embolism
Keywords: intermediate-high; acute pulmonary embolism; systemic thrombolysis; catheter- directed management
MeSH Terms: interventions — Streptokinase

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- patients who received systemic thrombolysis: patients have been diagnosed with acute intermediate-high pulmonary embolism received I.V. streptokinase if there are no contraindications.
  Interventions: Drug: Streptokinase Injection
- patients who underwent catheter-based intervention: patients have been diagnosed with acute intermediate-high pulmonary embolism underwent catheter-based intervention including thrombus aspiration or catheter directed thrombolysis using Penumbra System
  Interventions: Device: Penumbra System

INTERVENTIONS:
Drug: Streptokinase Injection — 250000 IU as a loading dose over 30 min. Followed by 100000 IU/hour over 12:24hours or accelerated regimen 1.5 million IU over 2 hours
  Other Names: Kabikinase; Streptase
  Groups: patients who received systemic thrombolysis
Device: Penumbra System — which comprised of several devices:
  * RED Reperfusion Catheters
  * Penumbra JET Reperfusion Catheters
  * ACE Reperfusion Catheters
  * MAX Reperfusion Catheters
  * 3D Revascularization Device
  * Penumbra ENGINE Aspiration Source
  * Penumbra ENGINE Canister
  * Aspiration Tubing
  Groups: patients who underwent catheter-based intervention

SUMMARY:
To compare in hospital clinical outcomes and one month follow up of systemic thrombolysis versus catheter directed management for the treatment of acute intermediate- high risk pulmonary embolism (using streptokinase or tissue plasminogen activator (TPA) and catheter-based intervention group using Penumbra System).

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with acute intermediate-high pulmonary embolism

Exclusion Criteria:

* Patients less than 18 years of age.
* Low risk, intermediate low risk, acute pulmonary embolism
* patients with RV masses will be excluded.
* Patient refusal of treatment strategy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be subjected to:
  On admission:
  Detailed history for assessment of risk factors
  Clinical examination:
  Laboratory investigations.
  Trans-thoracic echocardiography to detect signs of PE:
  MSCT pulmonary angiography: for assessment of site, size and shape of pulmonary embolism.
  PESI and sPESI scores will be calculated for all patients.
  In hospital follow up:
  During hospital stay all patients will be followed up daily for assessment of hemodynamic, oxygen saturation, TTE, troponin level, need of mechanical ventilation or death.
  One month follow up after discharge: for the assessment of:
  Hemodynamic. Transthoracic echocardiography. MSCT pulmonary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2029-11-30 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure | during hospital stay (about 1 week) and one month after discharge
Change in heart rate | during hospital stay (about 1 week) and one month after discharge
Change in respiratory rate | during hospital stay (about 1 week) and one month after discharge
Change of O2 saturation. | during hospital stay (about 1 week)
Change of RV signs of PE by Transthoracic echocardiography | during hospital stay (about 1 week) and one month after discharge
Need for mechanical ventilation. | during hospital stay (about 1 week)
Need for surgical intervention. | during hospital stay (about 1 week)
  surgical embolectomy
Duration of hospital stay. | during hospital stay (about 1 week)

SECONDARY OUTCOMES:
incidence of Perforation of pulmonary artery | during hospital stay (about 1 week)
  may occur during catheter directed interventions
incidence of pericardial effusion | during hospital stay (about 1 week) and one month after discharge
  due to: infection cardiac perforation during catheter directed interventions
incidence of Major bleeding | during hospital stay (about 1 week) and one month after discharge
  that requires blood transfusions or urgent intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ayman K Mohamed, PHD, Principal Investigator — Assiut University; Mohamed O Abdelhameed, master, Study Director — Assiut University
Locations (1):
- Hospital University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
compare in hospital clinical outcomes and one month follow up of systemic thrombolysis versus catheter directed management for the treatment of acute intermediate- high risk pulmonary embolism (using streptokinase or tissue plasminogen activator (TPA) and catheter-based intervention group using Penumbra System).
Supporting Information: Study Protocol, SAP, CSR